CLINICAL TRIAL: NCT06720545
Title: Cardiometabolic Risk Effects of Short-term Cessation of Effective Neurostimulation Therapy in OSA
Brief Title: Cardiometabolic Risk Effects of Short-term Cessation of Neurostimulation Therapy
Acronym: CRESCENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Academy of Sleep Medicine (Other); Triological Society (Unknown); American Heart Association (Other)
Responsible Party: Principal Investigator, Yi Cai, Director of Sleep Surgery, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU9827
Record Dates: First submitted 2024-10-01; First posted 2024-12-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea; Obstructive Sleep Apnea of Adult
Keywords: hypoglossal nerve stimulation; inspire
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Therapeutic HGNS (HGNS-on) (No Intervention): Prior to enrollment in this study, participants will have been implanted with and stabilized on HGNS therapy. As part of clinical care, a therapeutic voltage setting will have been confirmed via overnight sleep study. This arm of the study maintains the participants on the HGNS therapy at the therapeutic voltage they have been using. This is a representation of the patient's baseline status.
- No HGNS therapy (HGNS-off) (Other): HGNS therapy will be turned off by the participant for this arm of the study. This arm will mimic the participant's untreated OSA statement before they had HGNS therapy activated.
  Interventions: Device: No HGNS therapy (HGNS-off)

INTERVENTIONS:
Device: No HGNS therapy (HGNS-off) — Prior to enrollment in this study, participants will have been utilizing HGNS at a therapeutic voltage setting confirmed via overnight sleep study. As part of the trial, they will undergo a study arm that involves turning off HGNS therapy (HGNS-off) for between 2-4 weeks.
  Arms: No HGNS therapy (HGNS-off)

SUMMARY:
Hypoglossal nerve stimulation (HGNS) is an implantable therapy that treats obstructive sleep apnea.

The study will evaluate the effect of this treatment on cardiovascular and metabolism-related measures to see if it affects patients' risk of medical problems associated with obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults (18+ years) who have met surgical efficacy criteria with HGNS, as defined by at least a 50% reduction in apnea-hypopnea index (AHI) to <20 (with hypopneas defined by 4% oxyhemoglobin desaturations)
* Have been using HGNS therapy for at least 3 months and used HGNS for >20 hours/week during the past 4 weeks
* Were not using any OSA therapy for at least one month prior to HGNS activation or have had a one-month period of untreated OSA after HGNS activation

Exclusion Criteria:

* Chronic use of opiate medications, illicit drugs, or alcohol dependency
* Women who are pregnant or planning to become pregnant
* Shift workers, heavy machinery operators, or commercial drivers
* History of severe excessive daytime sleepiness (Epworth Sleepiness Scale score >16 at time of screening or prior to HGNS), motor vehicle accidents or near-miss incidents due to drowsy driving within the year prior to enrollment
* Significant cardiopulmonary (such as home oxygen requirement), liver, renal, or oncologic disease; neurodegenerative disease; active or recent history of an eating disorder (within the last 5 years)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Free living energy expenditure | Data will be obtained in the last 2 weeks of each study phase (HGNS-on or HGNS-off)
  The investigators will measure energy expenditure using the doubly labeled water (DLW) technique and actigraphy.
Hypoxic burden | Data will be obtained in the last 2 weeks of each study phase (HGNS-on or HGNS-off).
  The investigators will measure hypoxic burden based on the home sleep testing obtained during the study.

SECONDARY OUTCOMES:
Insulin resistance | These measures will be taken at the end of each study phase (duration of 2-4 weeks)
  Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) will be derived from fasting glucose and insulin

OTHER OUTCOMES:
Leptin levels | At the end of each study phase (duration of 2-4 weeks)
  Serum leptin will be measured using a double-antibody radioimmunoassay (RIA).
Adiponectin levels | At the end of each study phase (duration of 2-4 weeks)
  Adiponectin levels will be analyzed using RIA.
Ghrelin levels | At the end of each study phase (duration of 2-4 weeks)
  Total ghrelin will be assessed using RIA.
Glucagon-like peptide-1 (GLP-1) levels | At the end of each study phase (duration of 2-4 weeks)
  GLP-1 will be measured by RIA after plasma extraction with 95% ethanol.
E-selectin levels | At the end of each study phase (duration of 2-4 weeks)
  E-selectin will be measured as an inflammatory marker.
Vascular endothelial growth factor-A (VEGF-A) levels | At the end of each study phase (duration of 2-4 weeks)
  VEGF-A will be measured as an inflammatory marker.
Apnea-Hypopnea Index (AHI) | These measures will be taken at the end of each study phase (duration of 2-4 weeks)
  The participants will undergo home sleep testing, which will report an AHI value.
Height in meters | This measure will be taken at each study visit (duration of 1-4 weeks)
  Participants' height will be measured without shoes.
Weight in kilograms | This measure will be taken at every study visit (duration 1-4 weeks)
  Participants' weight will be measured after a urine void
Waist circumference in centimeters | This measure will be taken at every study visit (duration 1-4 weeks)
  Participants' waist circumference will be measured
Sleep duration (minutes) | Data will be obtained in the last 2 weeks of each study phase (HGNS-on or HGNS-off)
  The investigators will measure sleep duration in minutes based on actigraphy.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participant PHI protection